CLINICAL TRIAL: NCT02354573
Title: A Mechanistic Study to Assess The Role of Chronotropic Incompetence in Heart Failure With Normal Ejection Fraction (HFNEF)
Brief Title: The Role of Chronotropic Incompetence in Heart Failure With Normal Ejection Fraction (HFNEF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 11/SC/0009
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active arm (Active Comparator): All subjects will receive Ivabradine 7.5mg twice daily for 2 weeks in a double-blind randomized crossover design.
  Interventions: Drug: Ivabradine
- Placebo arm (Placebo Comparator): All subjects will receive matching placebo tablets twice daily for 2 weeks in a double-blind randomized crossover design.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — All subjects will receive Ivabradine 7.5mg twice daily for 2 weeks in a double-blind randomized crossover design.
  Other Names: Procoralan

SUMMARY:
What is heart failure with normal ejection fraction? The heart contracts (pumps) and relaxes with each heartbeat. In some people with heart failure, the heart contracts normally but there is reduced relaxation of the heart. As a result, people notice a feeling of breathlessness, ankle swelling and fatigue especially on exertion.

The investigators feel that patients with reduced or impaired relaxation of the heart have less heart filling time and poor energy utilisation during exercise. Therefore, the investigators are conducting a study to more thoroughly understand the disease condition by giving a drug called ivabradine to reduce the heart rate and hence to increase the heart filling time in these patients.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE About 50% of patients with heart failure have a normal ejection fraction (HFNEF). Although traditionally considered a more benign disorder than the related heart failure with reduced ejection fraction (HFREF), the mortality figures for patients with HFNEF and HFREF are now known to be comparable. Surprisingly, despite HFNEF's importance as a major health concern, the pathophysiological basis of HFNEF's remains poorly understood with some commentators even suggesting that HFNEF's pathophysiology is a variant of HFREF. Further confounding the understanding of HFNEF, existing studies included heterogenous patients of stratified ethnicities and ages who were assessed at rest. Such patients may not exhibit the same physiology as the typically elderly female HFNEF patients who experience symptoms during exertion.

Elucidating the mechanisms underlying HFNEF is pressing as there is a paucity of evidence to even begin to guide therapy. In the absence of supportive trial evidence, clinical practice has been predicated on assumptions made regarding the physiology of diastolic (dys)function. For example, rate limitation is often advocated in HFNEF based on the 19th century observations by Lewis Katz that at higher heart rates, shortening of diastolic filling period impairs cardiac filling and results in lower stroke volumes.

Such empirical practices are beset by HFNEF's complexity. A consistent feature of HFNEF is reduced chronotropic reserve. In one study HFNEF patients were assessed invasively using pressure-volume loops during basal conditions and handgrip exercise with atrial pacing at 120bpm. It was concluded that at higher heart rates, there was a significant blunting of frequency-dependent ventricular relaxation and that rate-related diastolic chamber stiffness compromised stroke volume explaining exertional limitation. Other investigators have disputed the aberrancy of diastolic filling limitation, questioning the potential benefits of heart rate limitation using beta-blockers and raising the potential for pacing as a treatment for HNEF. We confirmed the impaired chronotropic reserve in HFNEF. We also demonstrated dynamic slowing of LV relaxation during exercise that was associated with and potentially attributable to impaired cardiac energetics (albeit at rest)9. However, to determine the pertinence of heart rate to inadequate exertional reserve in HFNEF, heart rate needs to be manipulated in the complex neurohormonal, autonomic and haemodynamic context of exercise. The fundamental limitation of existing studies, including those utilizing pacing and handgrip, is that exercise physiology was not recapitulated.

Cardiac MR is the most accurate and versatile method for phenotyping the heart in research studies, and can assess cardiac volumes and mass with unparalleled accuracy and reproducibility. 31P MRS is the only technique that allows non-invasive measurement of cardiac high-energy phosphate metabolism in vivo. Our department has developed a 31P-MRS protocol which allows for measuring high energy phosphate molecules at rest and during exercise Cardiopulmonary exercise testing with peak oxygen consumption measurement has been shown to be a reliable mechanistic readout of integrated cardiac function in heart failure with preserved ejection fraction9,. It is also safe and reliable in elderly patients with heart failure.

In summary, chronotropic incompetence could either be a compensatory phenomenon serving to limit cardiac energetic depletion on exercise and also increasing diastolic filling in the context of an abbreviated diastolic filling time due to dynamic slowing of active relaxation. Alternatively it might contribute to exercise limitation by limiting cardiac output augmentation on exercise (since cardiac output is the product of heart rate and stroke volume). In order to investigate this LV filling and cardiac output pathophysiology in HFNEF, we will employ Ivabradine, that reduces heart rate but has no direct effect on contractile/lusitropic function or on vascular tone.

Ivabradine is indicated in symptomatic chronic stable angina patients who are unable to tolerate or with a contra-indication to the use of beta-blockers. It can be used in combination with beta-blockers whose heart rate is > 60 bpm. We will use ivabradine as a pharmacological tool to investigate diastolic filling/function and hence its effect on cardiac function and metabolism of energy. Ivabradine dose has been extensively validated and deemed safe in the a previous study (Beautiful study). The common side effects are transient enhanced brightness in a limited area of the visual field, usually triggered by sudden variations in light intensity and blurred vision. Other common side effects are bradycardia, headache and dizziness possibly related to bradycardia.

Ivabradine is metabolised by CYP3A4 and the concomitant use of potent CYP3A4 inhibitors such as azole antifungals (ketoconazole, itraconazole), macrolide antibiotics (clarithromycin, erythromycin, josamycin, telithromycin), HIV protease inhibitors and nefazodone is contraindicated. The combination of ivabradine with the heart rate reducing agents diltiazem or verapamil is not recommended. Other drugs which combination with ivabradine is not recommended are QT prolongation drugs (quinidine, disopyramide, bepridil, sotalol, ibutilide, amiodarone, pimozide, ziprasidone, sertindole, mefloquine, halofantrine, pentamidine). Combination of ivabradine with beta-blockers, ACE inhibitors, angiotensin II antagonists, diuretics, short and long acting nitrates, HMG CoA reductase inhibitors, fibrates, proton pump inhibitors, oral antidiabetics, aspirin, and other anti-platelet agents has been found to be safe.

Although not a clinical trial, we will assess the impact of lowering heart rate on exercise in patients with HFNEF and in matched patients with hypertension but no exercise limitation in order to begin to understand the role of heart rate in diastolic physiology.

Patient selection Through our HFNEF community screening programme, and via heart failure clinics in Oxford we will identify 30 patients with HFNEF who meet ESC criteria and additionally have peak VO2 ≤ 85% with a cardiac pattern of exercise limitation during CPEX; 30 matched hypertensive controls without HFNEF (no subjective complaint of breathlessness and peak V02 > 90% of age and gender predicted) will be recruited and studied in Aberdeen by a research team led by Professor Michael Frenneaux. 20 matched healthy subjects will be recruited in Oxford to provide normal reference values for study examinations at baseline.

STUDY DESIGN Summary of study design This research project has 3 groups and will be done in 2 different centres, Oxford and Aberdeen. Both HFNEF and hypertensive controls (positive controls) will participate in a prospective, randomized, double-blind, placebo-controlled crossover design consisting of two experimental periods (Ivabradine 7.5mg bd vs placebo each for two weeks with two weeks washout in between). Normal controls (negative controls) will only undergo baseline assessments and will not be given Ivabradine or placebo.

Group 1 (University of Oxford) This will be done by a research team led by Dr Houman Ashrafian and Prof S Neubauer.

30 patients with HFNEF, who are at least 60 years old will be recruited from the heart failure clinic at the John Radcliffe Hospital or the HFNEF community screening programme in Oxford over a 24-month period. Only those with VO2max of ≤ 85% with a cardiac pattern of exercise limitation during CPEX at screening will be included in the study.

At the end of screening visit, all eligible subjects will be randomly assigned to one of the possible experimental sequences. Each subject will receive either Ivabradine 7.5mg bd or matching placebo tablets (Period 1), followed by a 2-week washout period, and then placebo or Ivabradine 7.5mg bd for the final 2-week period (Period 2). The subject and study investigators will be blind to the randomization schedule. Patients will be evaluated at baseline and at the end of the two experimental periods in John Radcliffe hospital. All the evaluation days will last approximately 4 hours.

Elderly participants will be allowed to perform MRI/MRS on the next day.

Group 2 (University of Aberdeen) This will be done by a research team led by Professor Michael Frenneaux. 30 matched hypertensive controls, without heart failure symptoms who are at least 65 years old will be recruited in Aberdeen over a 24-month period. Only those with VO2max of > 90% predicted during CPEX at screening will be included in the study.

Elderly participants will be allowed to perform nuclear study or MRI/MRS on the next day.

Group 3 (Normal Subjects) 20 matched normal controls, who are at least 18 years old will be recruited in Oxford over a 24-month period. All participants will only undergo Visit 1 tests and will not be given Ivabradine or placebo.

Study Procedures Eligibility of patients will be checked by predefined inclusion/exclusion criteria at the time of attendance to the heart failure clinic (Oxford), cardiology clinics, cardiac investigation department and other relevant clinics in John Radcliffe hospital (such as hypertension, diabetes e.t.c.) or hypertension/cardiology clinic (Aberdeen Royal Infirmary) by the clinical team.

Informed Consent Written and verbal explanation of the study aims and protocol will be provided detailing the exact nature of the study, the implications and constraints of the protocol and the known possible side effects and any risks involved in taking part.

Study Assessments

Screening visit, 1-2 hours

1. Check for eligibility
2. Obtain written informed consent
3. History and physical examination
4. Cardiopulmonary exercise testing (CPEX)

   * VO2 max.
   * Ventilatory efficiency (VE/VCO2)
   * Respiratory exchange ratio
   * Lactate level (optional)

   Only those eligible [peak V02 ≤ 85% with a cardiac pattern of exercise limitation during CPX (Group 1, Oxford) or peak V02 > 90% (Group 2, Aberdeen)] will continue with rest of screening visit study procedures. Participants who are not eligible will be withdrawn from the study at this point.
5. To complete MLHFQ
6. Resting ECG
7. Bloods (10ml draw) for FBC, renal profile, fasting glucose, cholesterol, liver function, FFA and BNP.

At the end of screening visit, subjects will be randomly assigned to either Ivabradine 7.5mg twice daily or matching placebo tablets for 2 weeks (Period 1).

Visit 1 (4 hours, 2 weeks after starting Period 1 - Ivabradine/placebo) All assessments at screening will be repeated (barring seeking written consent again) and all experimental agents will be stopped. Additionally a cardiac MRI scan will be performed.

Visit 2 (4 hours, 2 weeks after starting Period 2 - placebo/Ivabradine) All visit 1 assessments will be repeated and all tablets will be stopped. All subjects will be requested to return all unused tablets from the Period 2. The study will end at the end of Visit 2.

Healthy volunteers (group 3) will only undergo all assessments as a single visit and will not undergo CPEX screening test or given a study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participant who is willing and able to give informed consent for participation in the study.
* Male or Female, aged 60 years and over (Group 1, Oxford).
* Patients diagnosed with HFNEF by ESC criteria and have peak V02 ≤ 85% with a cardiac pattern of exercise limitation during CPEX (Group 1, Oxford).
* Hypertensive controls aged 65 and over without HFNEF and with peak V02 > 90% (Group 2, Aberdeen)
* Able to perform exercise testing.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* LVEF <50%
* Inability to tolerate MRI scanning (claustrophobia, inability to lie flat)
* Contraindications to CMR imaging (implantable devices or other metal implants, internal cardioverter-defibrillator, cranial aneurysm clips, metallic ocular foreign bodies, hypersensitivity to gadolinium)
* Presence of other significant concomitant diseases such as ischaemic, valvular, pericardial heart disease or cardiomyopathy.
* Presence of asthma (contraindication to adenosine)
* Presence of 2nd or 3rd degree AV block (contraindications to ivabradine and adenosine)
* Presence of sick sinus syndrome
* Presence of atrial fibrillation
* Significant bradycardia (HR <60 per minute).
* Objective evidence of lung disease on formal lung function testing
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study
* Unable to perform exercise testing
* Patient who is in terminally ill or is inappropriate for medication
* Known hypersensitivity to Ivabradine or adenosine
* Significantly impaired renal function (eGFR<30ml/min)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in VO2max measured by CPEX | After 2 weeks of intervention

SECONDARY OUTCOMES:
Doppler derived E/e' | After 2 weeks of intervention
  ECHO derived parameter
BNP (Brain natriuretic peptide) | After 2 weeks of intervention
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | After 2 weeks of intervention
  Quality of life assessed by the MLHFQ.

CONTACTS AND LOCATIONS:
Overall Officials: Houman Ashrafian, MRCP, Principal Investigator — University of Oxford
Locations (1):
- Univesrtity of Oxford, John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Bhatia RS, Tu JV, Lee DS, Austin PC, Fang J, Haouzi A, Gong Y, Liu PP. Outcome of heart failure with preserved ejection fraction in a population-based study. N Engl J Med. 2006 Jul 20;355(3):260-9. doi: 10.1056/NEJMoa051530. PMID 16855266
- [Background] De Keulenaer GW, Brutsaert DL. The heart failure spectrum: time for a phenotype-oriented approach. Circulation. 2009 Jun 23;119(24):3044-6. doi: 10.1161/CIRCULATIONAHA.109.870006. Epub 2009 Jun 8. No abstract available. PMID 19506105
- [Background] Zile MR, Baicu CF, Gaasch WH. Diastolic heart failure--abnormalities in active relaxation and passive stiffness of the left ventricle. N Engl J Med. 2004 May 6;350(19):1953-9. doi: 10.1056/NEJMoa032566. PMID 15128895
- [Background] Westermann D, Kasner M, Steendijk P, Spillmann F, Riad A, Weitmann K, Hoffmann W, Poller W, Pauschinger M, Schultheiss HP, Tschope C. Role of left ventricular stiffness in heart failure with normal ejection fraction. Circulation. 2008 Apr 22;117(16):2051-60. doi: 10.1161/CIRCULATIONAHA.107.716886. Epub 2008 Apr 14. PMID 18413502
- [Background] Yip GW, Frenneaux M, Sanderson JE. Heart failure with a normal ejection fraction: new developments. Heart. 2009 Oct;95(19):1549-52. doi: 10.1136/hrt.2009.176222. Epub 2009 Jul 29. No abstract available. PMID 19643767
- [Background] Kindermann M, Reil JC, Pieske B, van Veldhuisen DJ, Bohm M. Heart failure with normal left ventricular ejection fraction: what is the evidence? Trends Cardiovasc Med. 2008 Nov;18(8):280-92. doi: 10.1016/j.tcm.2008.12.003. PMID 19345315
- [Background] Phan TT, Abozguia K, Nallur Shivu G, Mahadevan G, Ahmed I, Williams L, Dwivedi G, Patel K, Steendijk P, Ashrafian H, Henning A, Frenneaux M. Heart failure with preserved ejection fraction is characterized by dynamic impairment of active relaxation and contraction of the left ventricle on exercise and associated with myocardial energy deficiency. J Am Coll Cardiol. 2009 Jul 28;54(5):402-9. doi: 10.1016/j.jacc.2009.05.012. PMID 19628114
- [Background] Wachter R, Schmidt-Schweda S, Westermann D, Post H, Edelmann F, Kasner M, Luers C, Steendijk P, Hasenfuss G, Tschope C, Pieske B. Blunted frequency-dependent upregulation of cardiac output is related to impaired relaxation in diastolic heart failure. Eur Heart J. 2009 Dec;30(24):3027-36. doi: 10.1093/eurheartj/ehp341. PMID 19720638
- [Background] Bergstrom A, Andersson B, Edner M, Nylander E, Persson H, Dahlstrom U. Effect of carvedilol on diastolic function in patients with diastolic heart failure and preserved systolic function. Results of the Swedish Doppler-echocardiographic study (SWEDIC). Eur J Heart Fail. 2004 Jun;6(4):453-61. doi: 10.1016/j.ejheart.2004.02.003. PMID 15182771
- [Background] Liu CP, Ting CT, Lawrence W, Maughan WL, Chang MS, Kass DA. Diminished contractile response to increased heart rate in intact human left ventricular hypertrophy. Systolic versus diastolic determinants. Circulation. 1993 Oct;88(4 Pt 1):1893-906. doi: 10.1161/01.cir.88.4.1893. PMID 8403335
- [Background] Fox K, Ford I, Steg PG, Tendera M, Ferrari R; BEAUTIFUL Investigators. Ivabradine for patients with stable coronary artery disease and left-ventricular systolic dysfunction (BEAUTIFUL): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Sep 6;372(9641):807-16. doi: 10.1016/S0140-6736(08)61170-8. Epub 2008 Aug 29. PMID 18757088
- [Background] Shivu GN, Abozguia K, Phan TT, Ahmed I, Henning A, Frenneaux M. (31)P magnetic resonance spectroscopy to measure in vivo cardiac energetics in normal myocardium and hypertrophic cardiomyopathy: Experiences at 3T. Eur J Radiol. 2010 Feb;73(2):255-9. doi: 10.1016/j.ejrad.2008.10.018. Epub 2008 Dec 3. PMID 19056193
- [Background] Ommen SR, Nishimura RA, Appleton CP, Miller FA, Oh JK, Redfield MM, Tajik AJ. Clinical utility of Doppler echocardiography and tissue Doppler imaging in the estimation of left ventricular filling pressures: A comparative simultaneous Doppler-catheterization study. Circulation. 2000 Oct 10;102(15):1788-94. doi: 10.1161/01.cir.102.15.1788. PMID 11023933
- [Background] Pennell DJ, Sechtem UP, Higgins CB, Manning WJ, Pohost GM, Rademakers FE, van Rossum AC, Shaw LJ, Yucel EK; European Society of cardiology; Soceity for Cardiovascular Magnetic Resonance. Clinical indications for cardiovascular magnetic resonance (CMR): Consensus Panel report. J Cardiovasc Magn Reson. 2004;6(4):727-65. doi: 10.1081/jcmr-200038581. No abstract available. PMID 15646878
- [Background] Hudsmith LE, Neubauer S. Magnetic resonance spectroscopy in myocardial disease. JACC Cardiovasc Imaging. 2009 Jan;2(1):87-96. doi: 10.1016/j.jcmg.2008.08.005. PMID 19356540
- [Background] Scardovi AB, Coletta C, De Maria R, Perna S, Aspromonte N, Feola M, Rosso G, Greggi M, Ceci V. The cardiopulmonary exercise test is safe and reliable in elderly patients with chronic heart failure. J Cardiovasc Med (Hagerstown). 2007 Aug;8(8):608-12. doi: 10.2459/01.JCM.0000281698.53983.4e. PMID 17667032
- [Background] Bacharach SL, Green MV, Borer JS, Hyde JE, Farkas SP, Johnston GS. Left-ventricular peak ejection rate, filling rate, and ejection fraction--frame rate requirements at rest and exercise: concise communication. J Nucl Med. 1979 Mar;20(3):189-93. PMID 24180035
- [Derived] Pal N, Sivaswamy N, Mahmod M, Yavari A, Rudd A, Singh S, Dawson DK, Francis JM, Dwight JS, Watkins H, Neubauer S, Frenneaux M, Ashrafian H. Effect of Selective Heart Rate Slowing in Heart Failure With Preserved Ejection Fraction. Circulation. 2015 Nov 3;132(18):1719-25. doi: 10.1161/CIRCULATIONAHA.115.017119. Epub 2015 Sep 2. PMID 26338956